CLINICAL TRIAL: NCT02623218
Title: Translational Research Examining Acupuncture Treatment in Traumatic Brain Injury
Acronym: TREAT-TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AOMA Graduate School of Integrative Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AOMA-5510
Record Dates: First submitted 2015-12-03; First posted 2015-12-07 (Estimated); Results first posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; acupuncture; transcranial doppler ultrasound
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- TBI-ACUP (Experimental): This group will receive the standard of care plus acupuncture treatments during the acute 10-day phase following a diagnosed TBI.
  Interventions: Device: Acupuncture
- TBI-SHAM (Sham Comparator): This group will receive the standard of care plus sham acupuncture treatments during the acute 10-day phase following a diagnosed TBI.
  Interventions: Device: Sham Acupuncture
- C-ACUP (Active Comparator): This group of participants without TBI will receive one acupuncture treatment and serve as a healthy control group.
  Interventions: Device: Acupuncture
- C-SHAM (Sham Comparator): This group of participants will receive one sham acupuncture treatment and serve as a healthy sham comparator group.
  Interventions: Device: Sham Acupuncture
- C-EX (Active Comparator): This group of participants without TBI will receive one acupuncture treatment following 30-60 minutes of aerobic exercise, and serve as a healthy control group.
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — An acupuncture needle is a device intended to pierce the skin in the practice of acupuncture. The device consists of a solid, stainless steel needle. The device may have a handle attached to the needle to facilitate the delivery of acupuncture treatment.
  Arms: C-ACUP; C-EX; TBI-ACUP
Device: Sham Acupuncture — Sham acupuncture will be performed at the same locations as verum acupuncture. Streitberger sham acupuncture needles look like real acupuncture needles, and appear as though the skin is being penetrated during the insertion technique, however they do not pierce the skin.
  Other Names: Streitberger Needle
  Arms: C-SHAM; TBI-SHAM

SUMMARY:
The purpose of this study is to examine the effects of acupuncture on cerebral blood flow (CBF) and blood biomarkers during the acute 10-day window following traumatic brain injury, to determine if those changes correlate with changes in biomarkers of brain health, neuropsychological testing, and symptomatic presentation.

DETAILED DESCRIPTION:
The primary aim of this study is to examine the effects of acupuncture on brain function and cognition during the acute 10-day window following mild traumatic brain injury.

Traumatic brain injuries (TBI) affect an estimated 1.7 to 2.3 million Americans every year. As the clinical importance of managing those with TBI grows, it is essential that therapies to help in the recovery and management of post-concussion symptoms are identified. Currently, the number one recommended treatment strategy is physical and cognitive rest, followed by gradual return to daily activities and exercise.

Cerebral blood flow declines following TBI, and can remain in a depressed state for ongoing lengths of time. The cellular vulnerability and symptomatic presentation following TBI is likely due to the metabolic imbalance between decreased cerebral blood flow and increased demand for glucose and adenosine triphosphate production. Animal and human studies have shown that acupuncture at locations both locally on the head and neck, as well as distally on the arms, hands, legs, and feet, can increase cerebral blood flow through the left (L) and right (R) middle cerebral artery (MCA), internal carotid artery (ICA), and basilar artery (BA).

Acupuncture has a long history of use in the treatment of acute and chronic pain, headaches, migraines, nausea, anxiety, and sleep disorders, however, studies specific to the utilization of acupuncture in managing symptoms following TBI are lacking.

The investigators hypothesize that that acupuncture treatments may improve cerebral blood flow resulting in overall improvements in brain function and cognition following TBI. Acupuncture may provide a safe treatment to improve outcomes following a TBI, and increase the rate of recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50
* Documented TBI (for TBI-ACUP and TBI-SHAM arms)
* Visual acuity and hearing adequate for outcomes testing
* Fluency in English
* Ability to provide informed consent
* Acupuncture naïve

Exclusion Criteria:

* Significant polytrauma that may interfere with follow-up and outcome assessment
* Patients with major debilitating baseline mental health disorders that would interfere with the validity of outcome assessment due to TBI
* Patients on psychiatric hold
* Patients with major debilitating baseline neurological diseases impairing baseline awareness, cognition, or validity of outcome assessment due to TBI
* Significant history of pre-existing conditions that would interfere with the likelihood of follow-up and validity of outcome assessment due to TBI
* Pregnancy in female subjects
* Prisoners or patients in custody
* Current participation in an observational or intervention trial for TBI
* Non-English speakers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Finnell, ND, Principal Investigator — AOMA Graduate School of Integrative Medicine; Amy Moll, M.A.O.M., Study Director — AOMA Graduate School of Integrative Medicine
Locations (1):
- Healing Response Acupuncture & Integrative Medicine, Dallas, Texas, United States

REFERENCES:
- [Background] Byeon HS, Moon SK, Park SU, Jung WS, Park JM, Ko CN, Cho KH, Kim YS, Bae HS. Effects of GV20 acupuncture on cerebral blood flow velocity of middle cerebral artery and anterior cerebral artery territories, and CO2 reactivity during hypocapnia in normal subjects. J Altern Complement Med. 2011 Mar;17(3):219-24. doi: 10.1089/acm.2010.0232. Epub 2011 Feb 27. PMID 21417808
- [Background] Im JW, Moon SK, Jung WS, Cho KH, Kim YS, Park TH, Ko CN, Park JM, Park SU, Cho SY. Effects of acupuncture at GB20 on CO2 reactivity in the basilar and middle cerebral arteries during hypocapnia in healthy participants. J Altern Complement Med. 2014 Oct;20(10):764-70. doi: 10.1089/acm.2013.0240. Epub 2014 Sep 16. PMID 25226574
- [Background] An YS, Moon SK, Min IK, Kim DY. Changes in regional cerebral blood flow and glucose metabolism following electroacupuncture at LI 4 and LI 11 in normal volunteers. J Altern Complement Med. 2009 Oct;15(10):1075-81. doi: 10.1089/acm.2009.0257. PMID 19848545

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One enrolled participant did not meet eligibility criteria.
Period: Overall Study
Arm/Group | TBI-ACUP | TBI-SHAM | C-ACUP | C-SHAM | C-EX
Started | 5 | 4 | 4 | 4 | 4
Completed | 5 | 3 | 4 | 4 | 4
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TBI-ACUP | TBI-SHAM | C-ACUP | C-SHAM | C-EX | Total
Number analyzed (Participants) | 5 | 4 | 4 | 4 | 4 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 4 | 4 | 4 | 21
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 5 | 4 | 4 | 4 | 4 | 21
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 4 | 4 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Blood Flow Velocity in the Left (L) and Right (R) Middle Cerebral Artery (MCA), Internal Carotid Artery (ICA), and Basilar Artery (BA).
Description: Cerebral blood flow velocity was assessed at baseline, post-fight, and post-acupuncture in the TBI-ACUP arm.
  Cerebral blood flow velocity was assessed at baseline, post fight, and post-sham acupuncture in the TBI-SHAM arm.
  Cerebral blood flow velocity was assessed at baseline, post exercise, and post-acupuncture in the C-EX arm.
  Cerebral blood flow velocity was assessed at baseline, and post-acupuncture in the C-ACUP arm.
  Cerebral blood flow velocity was assessed at baseline, and post-sham acupuncture in the C-SHAM arm.
Time Frame: At baseline, post-fight, post-exercise (up to 5 hours from baseline), post acupuncture/post sham acupuncture (within 3 hours from baseline)
Population: 1 participant in the TBI-SHAM group did not complete the study
Measure: Mean (Standard Deviation); unit: ml/sec
Arm/Group | TBI-ACUP | TBI-SHAM | C-ACUP | C-SHAM | C-EX
Number analyzed (Participants) | 5 | 4 | 4 | 4 | 4
ml/sec
  Change in baseline to post-fight L MCA: number analyzed (Participants) | 5 | 3 | 0 | 0 | 0
  Change in baseline to post-fight L MCA | 3.2 (4.8) | 6.7 (10.5) |  |  |
  Change in baseline to post-fight in R MCA: number analyzed (Participants) | 5 | 3 | 0 | 0 | 0
  Change in baseline to post-fight in R MCA | 4 (6.0) | 12.7 (8.4) |  |  |
  Change in baseline to post-fight in L ICA: number analyzed (Participants) | 5 | 3 | 0 | 0 | 0
  Change in baseline to post-fight in L ICA | -0.4 (6.8) | 3 (1.6) |  |  |
  Change in baseline to post-fight in R ICA: number analyzed (Participants) | 5 | 3 | 0 | 0 | 0
  Change in baseline to post-fight in R ICA | 2.4 (3.1) | 2.3 (2.6) |  |  |
  Change in baseline to post-fight in BA: number analyzed (Participants) | 5 | 3 | 0 | 0 | 0
  Change in baseline to post-fight in BA | 2.0 (4.9) | 4 (3.7) |  |  |
  Change in post-fight to post-acup/sham in L MCA: number analyzed (Participants) | 5 | 3 | 0 | 0 | 0
  Change in post-fight to post-acup/sham in L MCA | -5.6 (5.1) | -9.0 (2.2) |  |  |
  Change in post-fight to post-acup/sham in R MCA: number analyzed (Participants) | 5 | 3 | 0 | 0 | 0
  Change in post-fight to post-acup/sham in R MCA | 1.0 (6.0) | -3.0 (4.1) |  |  |
  Change in post-fight to post-acup/sham in L ICA: number analyzed (Participants) | 5 | 3 | 0 | 0 | 0
  Change in post-fight to post-acup/sham in L ICA | -0.6 (2.2) | -7.3 (1.2) |  |  |
  Change in post-fight to post-acup/sham in R ICA: number analyzed (Participants) | 5 | 3 | 0 | 0 | 0
  Change in post-fight to post-acup/sham in R ICA | -3.0 (5.7) | -4.7 (3.8) |  |  |
  Change in post-fight to post-acup/sham in BA: number analyzed (Participants) | 5 | 3 | 0 | 0 | 0
  Change in post-fight to post-acup/sham in BA | 2.0 (3.3) | -1.0 (5.0) |  |  |
  Change in baseline to post-acup/sham in L MCA: number analyzed (Participants) | 5 | 3 | 4 | 4 | 4
  Change in baseline to post-acup/sham in L MCA | -2.0 (7.3) | -2.7 (9.0) | 7.3 (11.1) | -2.8 (4.4) | -5.8 (7.2)
  Change in baseline to post-acup/sham in R MCA: number analyzed (Participants) | 5 | 3 | 4 | 4 | 4
  Change in baseline to post-acup/sham in R MCA | 5.0 (2.7) | 9.7 (11.6) | 7.0 (8.7) | 5.0 (10.2) | -1.5 (2.3)
  Change in baseline to post-acup/sham in L ICA: number analyzed (Participants) | 5 | 3 | 4 | 4 | 4
  Change in baseline to post-acup/sham in L ICA | -1.4 (6.9) | -4.0 (2.2) | -2.3 (3.1) | 0.0 (1.9) | -2.8 (4.0)
  Change in baseline to post-acup/sham in R ICA: number analyzed (Participants) | 5 | 3 | 4 | 4 | 4
  Change in baseline to post-acup/sham in R ICA | -0.6 (5.0) | -2.3 (1.2) | -1.5 (7.3) | -3.0 (8.1) | -1.0 (1.6)
  Change in baseline to post-acup/sham in BA: number analyzed (Participants) | 5 | 3 | 4 | 4 | 4
  Change in baseline to post-acup/sham in BA | 4.0 (2.1) | 1.0 (4.3) | 6.5 (3.4) | 0.0 (7.9) | 2.3 (2.7)
  Change in post-exercise to post acup/sham in L MCA: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4
  Change in post-exercise to post acup/sham in L MCA |  |  |  |  | -3.5 (1.7)
  Change in post-exercise to post acup/sham in R MCA: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4
  Change in post-exercise to post acup/sham in R MCA |  |  |  |  | 1.0 (5.9)
  Change in post-exercise to post acup/sham in L ICA: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4
  Change in post-exercise to post acup/sham in L ICA |  |  |  |  | -2.3 (4.3)
  Change in post-exercise to post acup/sham in R ICA: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4
  Change in post-exercise to post acup/sham in R ICA |  |  |  |  | -1.5 (5.7)
  Change in post-exercise to post acup/sham in BA: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4
  Change in post-exercise to post acup/sham in BA |  |  |  |  | -0.5 (3.8)

2. Secondary Outcome: Changes in Hopkins Verbal Learning Test
Description: The Hopkins Verbal Learning Test consists of a 12-item word list, composed of four words from each of three semantic categories which the patient must learn over three trials. For each trial, the subject is instructed to listen carefully as the examiner reads the word list and attempt to memorize the words. The score for total recall is the sum of all the correctly-recalled words from each trial, ranging from 0 to 36, with higher scores indicating better recall and retention.
Time Frame: At baseline, post-fight, post-exercise, and post-acupuncture/sham acupuncture
Population: 1 participant in the TBI-SHAM group did not complete the study. Data were not collected for the "Post-Exercise Total Recall Raw" assessment for all groups, and not for "Post Acupuncture/sham Total Recall Raw" assessment in the "CACUP", "C-SHAM" and "C-EX" Arms/Groups.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TBI-ACUP | TBI-SHAM | C-ACUP | C-SHAM | C-EX
Number analyzed (Participants) | 5 | 3 | 4 | 4 | 4
Units on a scale
  Baseline Total Recall Raw | 20.6 (2.33) | 25.7 (2.87) | 25.7 (1.70) | 28.5 (3.5) | 29 (3.54)
  Post-Exercise Total Recall Raw: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Post Acupuncture/sham Total Recall Raw: number analyzed (Participants) | 5 | 3 | 0 | 0 | 0
  Post Acupuncture/sham Total Recall Raw | 27 (1.26) | 27.7 (1.25) |  |  |

3. Secondary Outcome: Rivermead Post-Concussion Survey
Description: The Rivermead Post-Concussion Symptoms Questionnaire (RPQ) is a 16-item survey that assesses the severity of the most common post-concussion symptoms on a scale of 0 to 4, with a total score range from 0 to 64 with 64 denoting the greatest symptom severity").
Time Frame: Post-fight, Post-Acupuncture/Sham - TBI-ACUP and TBI-SHAM groups only
Population: The groups with zero did not take this post-concussion survey because those participants were healthy controls who did not have a concussion.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TBI-ACUP | TBI-SHAM | C-ACUP | C-SHAM | C-EX
Number analyzed (Participants) | 5 | 3 | 0 | 0 | 0
Units on a scale
  Post-fight Rivermead | 8.4 (7.00) | 4 (2.94) |  |  |
  Post-acupuncture/sham Rivermea | 2.2 (3.92) | 1.7 (2.36) |  |  |

ADVERSE EVENTS:
Arm/Group | TBI-ACUP | TBI-SHAM | C-ACUP | C-SHAM | C-EX
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/4 | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes